CLINICAL TRIAL: NCT05877768
Title: PCD-CT Registry: Evaluation of Photon Counting Detector-CT Based Image Parameters in the Assessment and Quantification of Coronary Artery Disease (EPIPHANY)
Brief Title: Evaluation of PCD-CT Based Image Parameters in the Assessment and Quantification of Coronary Artery Disease
Acronym: EPIPHANY
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Mainz (Other)
Responsible Party: Principal Investigator, Tilman Emrich, Dr. med., University Medical Center Mainz
Other Study IDs: PCD-CT Registry
Record Dates: First submitted 2023-05-10; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease: Patients with suspected coronary artery disease and those with known coronary artery disease and the suspicion of progressive disease who undergo clinically indicated Coronary Computed Tomography Angiography on the Photon-Counting Detector CT will be enrolled after written consent. All data from the CT scan and potential additional investigations (e.g. invasive coronary angiographies) will be collected. There will be no additional investigations for the purpose of the study. After 1, 2 and 5 years, participants will be asked to answer a health questionaire.
  Interventions: Diagnostic Test: Photon Counting Detector Coronary Computed Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Photon Counting Detector Coronary Computed Tomography Angiography — Clinically indicated Photon Counting Detector Coronary Computed Tomography Angiography for the suspicion of coronary artery disease or the progression thereof.
  Other Names: Photon-Counting Detector CT (Naeotom Alpha, Siemens Healthineers)

SUMMARY:
The goal of this observational study is to learn about a new type of computed tomography (Photon-Counting Detector CT) in patients with coronary artery disease.

The main questions it aims to answer are:

* How good is the image quality for the new CT
* How accurate are measurements in the images of the new CT
* Is there a relationship between measurements in the images and the management of the disease (e.g. new medication or additional investigations)
* Is there a relationship between measurements in the images and the results of follow-up investigations
* Is there a relationship between measurements in the images and the patient outcome

Participants will undergo normal clinical assessment of coronary artery disease and all data from the CT scan and additional investigations will be collected. There will be no additional investigations for the purpose of the study. After 1, 2 and 5 years, participants will be asked to answer a health questionaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for a coronary computed tomography angiography (CCTA) for the suspicion of coronary artery disease or the progression thereof
* Written informed consent

Exclusion Criteria:

* Contraindications preventing the execution of the CCTA (e.g., pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population screened for inclusion criteria will be patients referred for CCTA for suspected coronary artery disease and those with known coronary artery disease and the suspicion of progressive disease.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2033-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | From inclusion to a maximum follow-up of 5 years
  Composite endpoint: major adverse cardiovascular event (MACE); defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke.

SECONDARY OUTCOMES:
Objective Image Noise of Photon-Counting Detector Coronary Computed Tomography Angiography (PCD-CCTA) | during the PCD-CCTA examination
  Image Noise of PCD-CCTA measured objectively using measurements of CT values (HU).
Objective Assessment of Noise-Power Spectra of PCD-CCTA | during the PCD-CCTA examination
  Image Noise of PCD-CCTA measured objectively using noise-power spectra (W/Hz).
Subjective Image Noise of PCD-CCTA | during the PCD-CCTA examination
  Image Noise of PCD-CCTA judged subjectively on a 5-point Likert scale.
Objective Vessel sharpness in PCD-CCTA | during the PCD-CCTA examination
  Vessel sharpness in PCD-CCTA measured objectively using the slope of fitted double sigmoid curves (1/mm)
Subjective Vessel sharpness in PCD-CCTA | during the PCD-CCTA examination
  Vessel sharpness in PCD-CCTA judged subjectively on a 5-point Likert scale.
Objective Image Quality in PCD-CCTA | during the PCD-CCTA examination
  Objective Image Quality in PCD-CCTA measured objectively by contrast-to-noise ratio (HU/HU)
Subjective Image Quality in PCD-CCTA | during the PCD-CCTA examination
  Subjective Image Quality in PCD-CCTA judged subjectively on a 5-point Likert scale.
Influence of BMI on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of Body Mass Index (BMI, kg/m^2) on image quality of the PCD-CCTA
Influence of biological sex on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of patients biological sex (male/female) on image quality of the PCD-CCTA
Influence of monoenergetic energy levels on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of monoenergetic energy levels (keV) on image quality of the PCD-CCTA
Influence of slice thickness of reconstruction on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of slice thickness of reconstruction (mm) on image quality of the PCD-CCTA
Influence of reconstruction kernel on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of reconstruction kernel (Bv/Br/Qr) on image quality of the PCD-CCTA
Influence of kernel sharpness level on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of kernel sharpness level (40-90) on image quality of the PCD-CCTA
Influence of radiation dose on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of radiation dose (mGy) on image quality of the PCD-CCTA
Influence of the patients heart rate on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of the patients maximum, minimum and average heart rate (1/min) on image quality of the PCD-CCTA
Influence of the acquisition type on image quality of the PCD-CCTA | during the PCD-CCTA examination
  Influence of the acquisition type (Sequential, Spiral, Ultra-High Resolution, Spectral) on image quality of the PCD-CCTA
Quantitative analysis of Coronary Calcium Scoring from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of Coronary Calcium volume (mm^3), mass (g) and resulting score according to the Agatston classification.
Analysis of Stenosis Classification from PCD-CCTA | during the PCD-CCTA examination
  Analysis of Coronary stenosis classification according to the Coronary Artery Disease-Reporting and Data System (CAD-RADS, 0-5, higher numbers indicating more severe stenosis).
Quantitative analysis of Coronary Diameter Stenoses from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of Coronary Diameter Stenoses (%) from PCD-CCTA
Quantitative analysis of Coronary Area Stenoses from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of Coronary Area Stenoses (%) from PCD-CCTA
Quantitative analysis of computed Fractional Flow Reserve from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of computed Fractional Flow Reserve (absolute number) from PCD-CCTA.
Quantitative analysis of myocardial density from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of myocardial density (HU) from PCD-CCTA.
Quantitative analysis of myocardial iodine content from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of myocardial iodine content (µg/cm^3) from PCD-CCTA.
Quantitative analysis of extracellular volume fraction from PCD-CCTA | during the PCD-CCTA examination
  Quantitative analysis of the extracellular volume fraction (%) from PCD-CCTA.
Influence of BMI on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of Body Mass Index (BMI, kg/m^2) on quantitative parameters of the PCD-CCTA
Influence of biological sex on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of patients biological sex (male/female) on quantitative parameters of the PCD-CCTA
Influence of monoenergetic energy levels on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of monoenergetic energy levels (keV) on quantitative parameters of the PCD-CCTA
Influence of slice thickness of reconstruction on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of slice thickness of reconstruction (mm) on quantitative parameters of the PCD-CCTA
Influence of reconstruction kernel on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of reconstruction kernel (Bv/Br/Qr) on quantitative parameters of the PCD-CCTA
Influence of kernel sharpness level on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of kernel sharpness level (40-90) on quantitative parameters of the PCD-CCTA
Influence of radiation dose on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of radiation dose (mGy) on quantitative parameters of the PCD-CCTA
Influence of the patients heart rate on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of the patients maximum, minimum and average heart rate (1/min) on quantitative parameters of the PCD-CCTA
Influence of the acquisition type on quantitative parameters of the PCD-CCTA | during the PCD-CCTA examination
  Influence of the acquisition type (Sequential, Spiral, Ultra-High Resolution, Spectral) on quantitative parameters of the PCD-CCTA
Rates of patients undergoing further cardiac diagnostics | 2 weeks after initial PCD-CCTA, 1-year follow-up, 2-year follow-up and final follow-up up to a max of 5 years
  Rates of patients undergoing further cardiac diagnostics, such as additional CT or Invasive Coronary Angiography (ICA), Electrocardiography (ECG), Exercise ECG, Echo, Stress Echo, Magnetic Resonance Imaging (MRI) within 3 months following PCD-CCTA (defined as: related to these tests) and more than 3 months after PCD-CCTA until follow-up (unrelated to these tests).
Rates of patients undergoing cardiac interventions | 2 weeks after initial PCD-CCTA, 1-year follow-up, 2-year follow-up and final follow-up up to a max of 5 years
  Cardiac interventions such as coronary revascularization by ICA, coronary artery bypass grafting (CABG), Valve replacement (operatively and interventional), other cardiothoracic surgeries, implantation of an cardioverter/defibrillator or cardiac resynchronization device, ablation, others
Correlation and agreement of quantitative measurements from PCD-CCTA with ICA | ICA within 3 months of initial PCD-CCTA
  Correlation and agreement of percent diameter stenosis quantification by PCD-CCTA in comparison to quantitative assessment from ICA.
Correlation and agreement of non-invasive Fractional Flow Reserve from PCD-CCTA with invasive Fractional Flow Reserve from ICA | ICA within 3 months of initial PCD-CCTA
  Correlation and agreement of non-invasively estimated Fractional Flow Reserve by Computed Tomography with invasive Fractional Flow Reserve
Correlation and agreement of Percent diameter stenosis measurement from PCD-CCTA with Fractional Flow Reserve from ICA | ICA within 3 months of initial PCD-CCTA
  Correlation and agreement of stenosis quantification by PCD-CCTA and invasive Fractional Flow Reserve.
Correlation and agreement of Plaque composition assessment from PCD-CCTA with intracoronary techniques | ICA within 3 months of initial PCD-CCTA
  Correlation and agreement of Plaque composition assessment from PCD-CCTA in comparison to intracoronary techniques such as optical coherence tomography (OCT) in patients who had both tests done.
Correlation of quantitative PCD-CCTA parameters with the results of additional imaging ischemia tests | Imaging ischemia tests within 3 months of initial PCD-CCTA
  Correlation of quantitative PCD-CCTA parameters with imaging ischemia tests in patients who had both PCD-CCTA and one of the following tests done: stress echo, stress Single Photon Emission Computed Tomography (SPECT), stress Positron Emission Tomography (PET), and stress MRI.
Correlation of quantitative PCD-CCTA parameters with the results of additional other imaging tests | Imaging tests within 3 months of initial PCD-CCTA
  Correlation of quantitative PCD-CCTA parameters with imaging tests in patients who had both PCD-CCTA and one of the following tests done: transthoracic echo, transesophageal echo, cardiac MRI.
Patient management | at baseline, 1-year follow-up, 2-year follow-up and final follow-up up to a max of 5 years
  Recommended and actually performed management based on PCD-CCTA
Analysis of occurrence in Major Adverse Cardiac Events in subgroups | at baseline, 1-year follow-up, 2-year follow-up and final follow-up up to a max of 5 years
  Composite outcome: Analysis of occurrence in MACE as a secondary outcome in following subgroups:
  CT plaque characteristic groups: high risk versus other plaques versus no plaques; Plaque burden groups: P1 vs. P2 vs. P3 vs. P4 according to the CAD-RADS 2.0 classification; Gender: male versus female; Age: occurrence of MACE in patient a) under 45 years, b) between 45 and 65 years and c) over 65 years; BMI: Patients with BMI a) under 25, b) between 25 and 30 and c) over 30;

CONTACTS AND LOCATIONS:
Overall Officials: Tilman Emrich, MD, Principal Investigator — University Medical Center Mainz
Locations (1):
- University Medical Center Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No